CLINICAL TRIAL: NCT01214564
Title: A Phase 2a, Multi-Centre, Open-Label Study to Evaluate the Safety and Efficacy of PEP005(Ingenol Mebutate) Gel, 0.05%, in Patients With Seborrhoeic Keratosis on Non-head Locations
Brief Title: Study to Evaluate the Safety and Efficacy of PEP005(Ingenol Mebutate) Gel, 0.05%, in Patients With Seborrhoeic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Responsible Party: Jacqueline Morley, Clinical Research Team Leader, Peplin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEP005-033
Record Dates: First submitted 2010-10-03; First posted 2010-10-05 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Seborrheic Keratosis
Keywords: PEP005; Peplin; Seborrhoeic Keratosis
MeSH Terms: conditions — Keratosis, Seborrheic; Keratosis, Actinic | interventions — 3-ingenyl angelate; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Up to three days of treatment
  Interventions: Drug: PEP005 (ingenol mebutate) Gel

INTERVENTIONS:
Drug: PEP005 (ingenol mebutate) Gel — 0.05%

SUMMARY:
This study is primarily designed to investigate whether treatment, once daily for up to three consecutive days, with PEP005 (ingenol mebutate) Gel, 0.05% will be safe and tolerable in patients with Seborrhoeic Keratosis on non-head locations. The secondary endpoint is to investigate the efficacy of PEP005 Gel, 0.05% when administered for up to three consecutive days to Seborrhoeic Keratosis on non-head locations.

ELIGIBILITY:
Inclusion Criteria

1. Patient is male or female and at least 18 years of age.
2. Female patients must be of either:

   * Non-childbearing potential, provided there is a laboratory confirmed serum follicle stimulating hormone (FSH) level ≥ 40mIU/ml or there is a confirmed clinical history of sterility (e.g., the patient is without a uterus); or
   * Childbearing potential, provided there are negative urine pregnancy test results prior to study treatment, to rule out pregnancy.
3. Patient has provided informed consent documented by signing the Informed Consent Form (ICF) prior to any study-related procedures, including any alteration of medications in preparation for study entry.
4. Patient has agreed to allow photographs of the selected treatment lesions to be taken and used as part of the study data package.

Exclusion Criteria

1. Known sensitivity or allergy to any of the ingredients in PEP005 (ingenol mebutate)Gel.
2. Current enrolment or participation in a clinical research study within 30 days of entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of PEP005 Gel, 0.05% when administered for up to three consecutive days to Seborrhoeic Keratosis on non-head locations. | Day 43

SECONDARY OUTCOMES:
To determine the efficacy of PEP005 Gel, 0.05% when administered for up to three consecutive days to Seborrhoeic Keratosis on non-head locations. | Day 43

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Southderm Pty Ltd, Kogarah, New South Wales
  - Specialist Connect, Woolloongabba, Queensland

REFERENCES:
- See also: Related Info — http://www.tga.gov.au/